CLINICAL TRIAL: NCT02414672
Title: CareSTEPS: A Supportive Care Program for the Caregivers of Advanced Lung Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Hoda Badr, Hoda Badr, PhD, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-38998; R01CA187143 (NIH)
Record Dates: First submitted 2015-04-07; First posted 2015-04-13 (Estimated); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Lung Cancer
Keywords: psychosocial intervention; advanced lung cancer; caregivers; self-care
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CareSTEPS (Experimental): CareSTEPS provides skills training in six domains that are central to the caregiving role: self-care, stress management, symptom management, effective communication, problem-solving, and social support.
  Interventions: Behavioral: CareSTEPS
- Usual Medical Care (UMC) (No Intervention): Patients receive standard oncologic and generalist palliative care from their healthcare team.

INTERVENTIONS:
Behavioral: CareSTEPS — Caregivers receive a workbook and 6 one-hour telephone sessions with a trained interventionist.
  Arms: CareSTEPS

SUMMARY:
The CareSTEPS intervention fills an important service gap by providing education, skills training, and support to the caregivers of advanced lung cancer patients on active treatment. The home-based delivery format will facilitate future dissemination and outreach. By empowering families with the skills they need to provide care and meet the challenges of lung cancer, this intervention holds great promise for improving caregiver quality of life (QOL), patient QOL, and the quality of palliative and supportive care services offered to patients with advanced cancer and their families.

DETAILED DESCRIPTION:
The profound symptom burden associated with advanced lung cancer (LC) makes caregiving a complex and burdensome task. Despite the input of outpatient palliative care services, LC families are often unprepared for caregiving, have low self-efficacy for managing symptoms at home, report high rates of physical and emotional distress, and receive very little skills training or psychosocial care. To date, the few psychosocial intervention trials targeting the caregivers of advanced cancer patients that have been conducted have mostly targeted the families of hospice patients, have not been well-integrated into routine palliative care, and have not addressed the specific needs of LC caregivers. Based on our published and recently completed pilot work in LC, the investigators have developed a psychosocial intervention called CareSTEPS (self-Care, Stress management, sympTom management, Effective communication, Problem-solving, and Social support). CareSTEPS is grounded by Self Determination Theory (SDT) which focuses on individuals' needs for developing autonomy (a sense of choice and volition), competence (self-efficacy), and relatedness (a sense of belonging and connection). It: 1) teaches skills to enhance caregiver competence for managing symptoms, practicing self-care, and coping with cancer; 2) supports caregiver autonomy by providing a clear rationale for recommendations and a variety of options to encourage choice and elaboration; and, 3) seeks to improve caregivers' sense of relatedness by teaching strategies for effective communication and soliciting/accepting social support. 200 LC patients will be enrolled within one month of treatment initiation (baseline) and their caregivers and randomize them to either a usual medical care (UMC) condition or the CareSTEPS intervention (caregivers receive a manual and six 45-minute weekly counseling sessions by telephone). The primary aim is to determine the impact of the CareSTEPS intervention on caregiver self-care behaviors, physical and emotional QOL, and satisfaction with care. Secondary aims are to: 1a) examine the effects of CareSTEPS on the SDT constructs of competence, autonomy, and relatedness; 1b) test whether caregiver competence, autonomy and relatedness mediate the effects of CareSTEPS on caregiver outcomes as hypothesized; 2) explore whether sociodemographic, medical, and relationship factors moderate the effects of the CareSTEPS intervention on SDT constructs; and, 3) explore the effects of CareSTEPS on patient QOL, palliative care utilization, and satisfaction with care. CareSTEPS fills an important service gap by providing education, skills training, and support to the caregivers of advanced LC patients who are on active treatment. The home-based delivery format will facilitate future dissemination and outreach. By empowering families with the skills they need to provide care and meet the challenges of LC, CareSTEPS holds great promise for improving caregiver QOL, patient QOL, and the quality of palliative/supportive care services for advanced cancer patients and their families.

ELIGIBILITY:
Inclusion Criteria:

* Patient has stage 3B or 4 NSLC or extensive stage SCLC and is within one month of treatment initiation
* Patient is spending more than 50% of time out of bed on a daily basis, as measured by an ECOG Performance Status rating of level 0, 1, or 2
* Patient has a spouse/partner other or close family member who he/she defines as the primary caregiver
* Patient and caregiver > 18 years
* Patient/caregiver has the ability to read and understand English at a sixth grade level, as determined by his/her ability to understand the consent form
* Patient/caregiver can provide informed consent

Exclusion Criteria:

* Individuals with diminished mental capacity
* Prisoners
* Children
* Pregnant Women
* Fetuses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Caregiver Depression | 8 weeks
  PROMIS Depression Short Form
Caregiver Anxiety | 8 weeks
  PROMS Anxiety Short form

SECONDARY OUTCOMES:
Caregiver burden | 8 weeks and 6 months
  Zarit Burden Interview
Patient emotional quality of life | 8 weeks and 6 months
  PROMIS Depression and Anxiety Short Forms
Caregiver Depression | 6 months
  PROMIS Depression Short Form
Caregiver Anxiety | 6 months
  PROMIS Anxiety Short Form

OTHER OUTCOMES:
Patient physical quality of life | 8 weeks and 6 months
  MD Anderson Symptom Inventory (MDASI-LC)
Caregiver Self-care behaviors | 8 weeks and 6 months
  Self-Management Behaviors (based on Lorig, 1996) Self-care (based on Schulz, 1999)
Caregiver Satisfaction with Care | 8 weeks and 6 months
  FAMCARE Scale
Caregiver physical quality of life | 8 weeks and 6 months
  Physical summary scale of the Short Form 12 (SF12)

CONTACTS AND LOCATIONS:
Overall Officials: Hoda Badr, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Rangel ML, Milbury K, Kayser K, Ripley RT, Kvale E, Badr H. Multisite Randomized Controlled Trial of CareSTEPS: A Supportive Care Intervention for the Family Caregivers of Patients With Advanced Lung Cancer. JTO Clin Res Rep. 2024 Oct 17;5(12):100736. doi: 10.1016/j.jtocrr.2024.100736. eCollection 2024 Dec. PMID 39583146